CLINICAL TRIAL: NCT00021827
Title: Pathophysiology of PTH-related Protein in Humans.
Brief Title: PTHrP and Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: PTHrP and Osteo (completed); RO-1 DK 51081
Record Dates: First submitted 2001-08-04; First posted 2001-08-06 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Osteoporosis
Keywords: parathyroid hormone-related protein; parathyroid hormone; anabolic skeletal therapy; postmenopausal women
MeSH Terms: conditions — Osteoporosis | interventions — Parathyroid Hormone-Related Protein

INTERVENTIONS:
Drug: Parathyroid hormone-related protein or ''PTHrP''

SUMMARY:
PTH-related protein, or ''PTHrP'', is a hormone which was discovered in 1987. As its name implies, it is closely related to another hormone discovered in the 1920's named parathyroid hormone or ''PTH''. PTH has been shown to be effective in treating osteoporosis in both animals and humans. PTHrP has been shown to be effective in treating osteoporosis in laboratory animals, and there are strong scientific reasons to think that it may be effective in humans as well. However, no human trials with PTHrP in the treatment of osteoporosis have been performed. The studies in this trial are focussed on determining whether PTHrP can indeed increase bone mass in postmenopausal women with osteoporosis, when administered daily by subcutaneous injection for three months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy caucasian postmenopausal females between 50-75 years of age with low bone mineral density at the lumbar spine or hip as measured using dual energy x-ray absorptiometry or DXA.
* ON estrogen replacement treatment for at least three years.

Exclusion Criteria:

* Heart, vascular, kidney, liver, lung, hormonal, musculo-skeletal disease (other than osteoporosis), rheumatic, blood diseases are exclusion criteria.
* High blood pressure
* Pregnancy
* Cancer
* Alcohol or drug dependence
* Prior use of a drug treatment for osteoporosis such as PTH, bisphosphonates, raloxifene, or calcitonin within the preceding five years

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-06; Study Completion 2001-12

CONTACTS AND LOCATIONS:
Overall Officials: Andrew F. Stewart, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Plotkin H, Gundberg C, Mitnick M, Stewart AF. Dissociation of bone formation from resorption during 2-week treatment with human parathyroid hormone-related peptide-(1-36) in humans: potential as an anabolic therapy for osteoporosis. J Clin Endocrinol Metab. 1998 Aug;83(8):2786-91. doi: 10.1210/jcem.83.8.5047. PMID 9709948
- [Background] Stewart AF, Cain RL, Burr DB, Jacob D, Turner CH, Hock JM. Six-month daily administration of parathyroid hormone and parathyroid hormone-related protein peptides to adult ovariectomized rats markedly enhances bone mass and biomechanical properties: a comparison of human parathyroid hormone 1-34, parathyroid hormone-related protein 1-36, and SDZ-parathyroid hormone 893. J Bone Miner Res. 2000 Aug;15(8):1517-25. doi: 10.1359/jbmr.2000.15.8.1517. PMID 10934650
- [Background] Syed MA, Horwitz MJ, Tedesco MB, Garcia-Ocana A, Wisniewski SR, Stewart AF. Parathyroid hormone-related protein-(1--36) stimulates renal tubular calcium reabsorption in normal human volunteers: implications for the pathogenesis of humoral hypercalcemia of malignancy. J Clin Endocrinol Metab. 2001 Apr;86(4):1525-31. doi: 10.1210/jcem.86.4.7406. PMID 11297578